CLINICAL TRIAL: NCT00104624
Title: Phase II Trial Assessing the Impact on Instrumental and Daily Living Autonomy of a Chemotherapy With Biweekly Docetaxel in the Treatment of Metastatic Breast Cancer in Patients Over 70
Brief Title: Docetaxel in Treating Older Women With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxicity issues
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000417747; FRE-FNCLCC-GERICO-04/0406; EU-20504
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well docetaxel works in treating older women with metastatic breast cancer and whether it helps improve the ability to perform daily activities.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine degree of autonomy in instrumental activities of daily living on-therapy and at 6 and 12 months, as measured by Lawton's Instrumental Activities of Daily Living Scale, in older women with metastatic adenocarcinoma of the breast treated with docetaxel.

Secondary

* Determine the response rate in patients treated with this drug.
* Determine overall and progression-free survival of patients treated with this drug.
* Determine the degree of autonomy in daily activities as measured by Katz's Activities of Daily Living Scale, in patients treated with this drug.
* Determine mood status, as measured by the Geriatric Depression Scale, of patients treated with this drug.
* Determine toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV on days 1 and 15. Treatment repeats every 28 days for 6 courses.

Ability to perform daily activities is assessed periodically.

PROJECTED ACCRUAL: A total of 53 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Metastatic disease
* Measurable disease by CT scan or MRI
* Requires first-line chemotherapy for metastatic disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 70 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Meets both of the following criteria:

  * Lawton's Instrumental Activities of Daily Living score ≥ 4
  * Katz's Activities of Daily Living score ≥ 4

Life expectancy

* More than 3 months

Hematopoietic

* Hemoglobin > 10 g/dL
* Neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* ALT and AST < 1.5 times normal
* Bilirubin normal
* Alkaline phosphatase < 2.5 times normal

Renal

* Creatinine clearance > 30 mL/min

Cardiovascular

* No congestive heart failure
* No unstable angina pectoris
* No myocardial infarction within the past year
* No uncontrolled hypertension
* No high-risk uncontrolled arrhythmias

Other

* Geriatric Depression Score < 12
* No active uncontrolled infection
* No active peptic ulcer
* No uncontrolled diabetes mellitus
* No inflammatory bowel disease
* No history of hypersensitivity to docetaxel or drugs formulated with polysorbate 80
* No history of significant neurologic or psychiatric disorders, including psychotic disorders, dementia, or seizures, that would preclude giving informed consent
* No familial, social, geographical, or psychological condition that would preclude study follow-up
* No definite contraindication to corticosteroids
* No other serious illness or medical condition
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior or concurrent trastuzumab (Herceptin^®)

Chemotherapy

* Prior neoadjuvant or adjuvant chemotherapy for breast cancer allowed
* More than 2 years since prior docetaxel or paclitaxel
* No other concurrent chemotherapy

Endocrine therapy

* No more than 1 prior hormonal therapy regimen for metastatic disease
* At least 10 days since prior hormonal therapy
* No concurrent hormonal therapy
* No concurrent chronic corticosteroids

  * Concurrent low-dose corticosteroids (≤ 20 mg/day of methylprednisolone or equivalent) allowed provided treatment was initiated > 6 months before study entry

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 30 days since prior active treatment on another clinical trial
* Concurrent bisphosphonates allowed for bone metastases, osteoporosis, or osteopenia
* No other concurrent anticancer therapy
* No other concurrent investigational drugs

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Degree of autonomy in instrumental activities of daily living as measured by Lawton's Instrumental Activities of Daily Living Scale during therapy and at 6 and 12 months

SECONDARY OUTCOMES:
Response rate
Overall survival
Degree of autonomy in daily activities as measured by Katz's Activities of Daily Living Scale
Progression-free survival
Mood status as measured by the Geriatric Depression Scale
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Delaloge, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (7):
- France (5):
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Institut Curie Hopital, Paris
  - Centre Henri Becquerel, Rouen
  - C.H. Senlis, Senlis
  - Institut Gustave Roussy, Villejuif
- Istituto Nazionale Di Riposo e Cura per Anziani, Rome, Italy
- Clinique De Genolier, Genolier, Switzerland